CLINICAL TRIAL: NCT01285791
Title: Sonographic Evaluation of Visceral and Subcutaneous Fat in Morbidly Obese Patients Before and After 3 Different Types of Bariatric Surgery.
Brief Title: Sonographic Evaluation of Visceral Fat After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ido Mizrahi, Ido Mizrahi MD, Hadassah Medical Organization
Other Study IDs: obesity17-HMO-CTIL
Record Dates: First submitted 2011-01-10; First posted 2011-01-28 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; intra-abdominal visceral fat; gastric bypass; sleeve gastrectomy; gastric banding; visceral fat
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients undergoing laparoscopic adjustable gastric banding: morbid obese patients undergoing laparoscopic adjustable gastric banding will be evaluated by ultrasound before surgery and one year after surgery to determine the amount of visceral fat layer decreased.
- patients undergoing laparoscopic sleeve gastrectomy: morbid obese patients undergoing laparoscopic sleeve gastrectomy will be evaluated by ultrasound before surgery and one year after surgery to determine the amount of visceral fat layer decreased
- patients undergoing laparoscopic gastric bypass: morbid obese patients undergoing laparoscopic gastric bypass will be evaluated by ultrasound before surgery and one year after surgery to determine the amount of visceral fat layer decreased

SUMMARY:
Excess visceral fat is a key factor in the development of metabolic syndrome associated with obesity. After bariatric surgery, patients experience weight loss accompanied by a decrease in the amount of total body fat. It is unclear how the different surgical procedures vary in their effect on the visceral and subcutaneous fat change. Ultrasonography (US) is an effective, efficient method in assessing this metabolically active layer of fat even when compared with gold standard techniques such as computed tomography and magnetic resonance imaging. Only a few studies managed to show the actual decrease in the visceral fat layer after these kinds of surgeries. The aim is to compare by ultrasound evaluation the extent of fat layers reduction after laparoscopic adjustable gastric banding (LAGB), laparoscopic sleeve gastrectomy (LSG) and laparoscopic roux-en-y gastric bypass (LRYGB). The hypothesis is that the sleeve gastrectomy and gastric bypass being not only a restrictive procedure but also a malabsorptive procedure will have the best results in decreasing the amount of visceral fat.

DETAILED DESCRIPTION:
excess visceral fat is a key factor in the development of metabolic syndrome associated with obesity. After bariatric surgery, patients experience weight loss accompanied by a decrease in the amount of total body fat. It is unclear how the different surgical procedures vary in their effect in reducing the amount of the visceral fat layer . Ultrasonography (US) is an effective, efficient method in assessing this metabolically active layer of fat even when compared with gold standard techniques such as computed tomography and magnetic resonance imaging. Only a few studies managed to show the actual decrease in the visceral fat layer after these kinds of bariatric surgeries. The aim is to compare by ultrasound evaluation the extent of fat layers reduction after laparoscopic adjustable gastric banding (LAGB), laparoscopic sleeve gastrectomy (LSG) and laparoscopic roux-en-y gastric bypass (LRYGB).

Visceral fat (VF) will be defined as the depth, in centimeters, from the rectus abdominis muscle to the aorta; and subcutaneous fat (SCF) defined as the depth, in centimeters, from the skin to the rectus abdominis muscle. Results will be compared with anthropometric measures as weight and waist circumference as well as laboratory results to try and find correlation between sonographic improvement and anthropometric and laboratory improvement.

The hypothesis is that the sleeve gastrectomy and gastric bypass being not only a restrictive procedure but also a malabsorptive procedure will have the best results in decreasing the amount of visceral fat.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years and below 70 years
* patients considered to suffer from morbid obesity as defined as a body mass index above 40 kg/meter*meter or above 35 kg/meter*meter with comorbidities relevant to obesity such as : diabetes, hypertension, arthralgia, obstructive sleep apnea and hyperlipidemia and eligible for surgery
* patients that electively and independently chose to undergo a bariatric surgery in our surgery ward.
* patients expressing their desire to participate in the study and after signing informed consent.
* patients that underwent a lecture about the pros and cons of the different types of bariatric surgery performed in our surgery ward:laparoscopic adjustable gastric banding, a sleeve gastrectomy or a gastric bypass and chose independently the type of surgery they want to undergo.
* patients that tried to lose weight in conventional ways such as physical activity and diets with no success.

Exclusion Criteria:

* patients under the age of 18 or above the age 70.
* patients unable to read, understand, comprehend and sign the informed consent form.
* patients not meeting the criteria for the definition morbid obesity as defined as a body mass index above 40 kg/meter*meter or above 35 kg/meter*meter with comorbidities relevant to obesity such as : diabetes, hypertension, arthralgia, obstructive sleep apnea and hyperlipidemia.
* pregnant patients.
* patients addicted to alcohol or other recreational drugs.
* patients suffering from a malignant comorbidity.
* patients suffering for a morbid obesity state because of a endocrine problem such as hypothyroidism or cushing disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbid obese patients admitted electively to our surgery ward after receiving detailed explanation about each type of surgery and after independently choosing to undergo either a laparoscopic adjustable gastric banding, a sleeve gastrectomy or a gatsric bypass will be offered to participate in the study.
  The patients must meet criteria for being morbid obese as defined as a body mass index greater than 40 kg/meter*meter or a body mass index greater than 35 with relevant comorbidities. The patients must meet other inclusion and exclusion criteria as defined below.
  The patients will be offered to participate in the study regardless of their gender or race.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ido Mizrahi, M.D, Principal Investigator — Ministry of Health, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
not planning on sharing data

REFERENCES:
- [Background] Del Genio F, Del Genio G, De Sio I, Marra M, Alfonsi L, Finelli C, Contaldo F, Pasanisi F. Noninvasive evaluation of abdominal fat and liver changes following progressive weight loss in severely obese patients treated with laparoscopic gastric bypass. Obes Surg. 2009 Dec;19(12):1664-71. doi: 10.1007/s11695-009-9891-x. PMID 19526270

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Undergoing Laparoscopic Adjustable Gastric Banding | Patients Undergoing Laparoscopic Sleeve Gastrectomy | Patients Undergoing Laparoscopic Gastric Bypass
Started | 11 | 15 | 13
Completed | 11 | 15 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Undergoing Laparoscopic Adjustable Gastric Banding | Patients Undergoing Laparoscopic Sleeve Gastrectomy | Patients Undergoing Laparoscopic Gastric Bypass | Total
Number analyzed (Participants) | 11 | 15 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (1.6) | 36.5 (3.1) | 38.7 (3) | 37.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 10 | 24
  Male | 4 | 8 | 3 | 15
Region of Enrollment [Number; unit: participants]
  Israel | 11 | 15 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Decrease in the Visceral Fat Layer Measured by Ultrasound a Day Before and a Year After Surgery.
Description: morbid obese patients undergoing a type of bariatric surgery either a laparoscopic gastric banding, a laparoscopic sleeve astrectomy or a laparoscopic gastric bypass, in our department will be evaluated by ultrasound 1 day before surgery and one year after surgery to determine the amount of visceral fat layer-by centimeters- that was decreased .
Time Frame: 18 months
Measure: Mean (Standard Error); unit: visceral fat reduction in centimeters
Arm/Group | Patients Undergoing Laparoscopic Adjustable Gastric Banding | Patients Undergoing Laparoscopic Sleeve Gastrectomy | Patients Undergoing Laparoscopic Gastric Bypass
Number analyzed (Participants) | 11 | 15 | 13
visceral fat reduction in centimeters | 3.6 (0.8) | 7.1 (0.5) | 5.6 (0.6)

2. Secondary Outcome: Change in Glucose and Triglyceride Blood Level
Description: finding correlation between sonographic outcome using ultrasound, as measured by the decrease in the level of visceral fat-by centimeters, weight loss and blood levels of triglycerides and glucose.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Patients Undergoing Laparoscopic Adjustable Gastric Banding | Patients Undergoing Laparoscopic Sleeve Gastrectomy | Patients Undergoing Laparoscopic Gastric Bypass
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes